CLINICAL TRIAL: NCT01760967
Title: Effect of Dexmedetomidine on Mortality, Duration of Mechanical Ventilation and Multi-organ Function in Sepsis Patients Under Lighter Sedation by Randomized Control Trial
Brief Title: Dexmedetomidine for Sepsis in ICU Randomized Evaluation Trial
Acronym: DESIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Collaborators: Osaka City University (Other); Hyogo Medical University (Other); Osaka City General Hospital (Other); National Hospital Organization Kyoto Medical Center (Unknown); Saga University (Other); Yamaguchi Grand Medical Center (Unknown); Sapporo Medical University (Other); Tohoku University (Other); Hirosaki University (Other); Kyoto Medical Center (Unknown)
Responsible Party: Principal Investigator, Yu Kawazoe, Assistant Professor, Tohoku University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DESIRE; UMIN000009665 (Other: UMIN-CTR)
Record Dates: First submitted 2012-12-26; First posted 2013-01-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Sepsis
Keywords: Dexmedetomidine; sepsis; mortality; duration of mechanical ventilation; organ failure
MeSH Terms: conditions — Sepsis | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): administer dexmedetomidine (0.1-0.7ug/kg/h) from the beginning of ICU treatment
  Interventions: Drug: Dexmedetomidine
- non-Dexmedetomidine (Active Comparator): administer sedatives except Dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — intervention to administer dexmedetomidine or not

SUMMARY:
Background:

Dexmedetomidine, a highly selective arfa2-adrenergic agonist, is known to be a unique sedative agent which causes less acute tolerance, drug addiction and withdrawal compared with gamma-aminobutyrate (GABA) agonists. Dexmedetomidine was approved for short-term ICU sedation in 2004 in Japan, and it has been used particularly for surgical ICU patients. In August 2010 dexmedetomidine was approved in Japan for sedation lasting more than 24 hours.

Recent evidence demonstrated that dexmedetomidine has organ protective effects including neuroprotection, cardioprotection, renal protection, gastrointestinal tract action, and anti-inflammatory action. Dexmedetomidine was shown to significantly decrease the infarct size in isolated rat hearts. Additionally, dexmedetomidine exhibited a preconditioning effect against ischemic injury in hippocampal slices, and this result was considered an apoptosis suppression effect of dexmedetomidine. Aydin C et al reported that dexmedetomidine enhanced the spontaneous contractions of the ileum in peritonitis rats compared with propofol and midazolam. Taniguchi and colleagues demonstrated that dexmedetomidine reduced high mortality rates and the plasma cytokine concentrations, interleukin-6 and tumor necrosis factor alpha in endotoxemic rats.

A meta-analysis has shown that perioperative alfa2-adrenergic agonists, including dexmedetomidine infusion, decreased cardiovascular events on patients undergoing cardiac surgery. Dexmedetomidine treated patients undergoing thoracotomy indicated increase in urine output, reduction in serum creatinine, and the suppression of diuretics in a randomized placebo-controlled double-blind study. Septic patients receiving dexmedetomidine had improved 28-day mortality rates compared with septic patients receiving lorazepam in a sub-group analysis of MENDS randomized controlled trial.

These positive effects of dexmedetomidine on the cardiovascular system, neurons, kidneys, gastrointestinal tract action, and an anti-inflammatory action, are expected to improve mortality in septic patients. However, large clinical research studies have not been conducted yet. We designed and conducted the DESIRE trial (DExmedetomidine for Sepsis in ICU Randomized Evaluation trial) to test a hypothesis that dexmedetomidine may improve clinical outcome and has these organ protective effects on septic patients.

Objective:

To determine whether dexmedetomidine improves clinical outcome and has organ protective effects on septic patients.

ELIGIBILITY:
Inclusion Criteria:

* adult
* transferred to ICU
* anticipation of a need for mechanical ventilation at least 24 hours

Exclusion Criteria:

* sever chronic liver disease (Child B or C)
* acute myocardial infarction, heart disease (NYHA 4)
* Drug dependence, alcoholism
* Psychological illness, severe cognitive dysfunction
* patients who have allergy for dexmedetomidine
* attending physician's decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
mortality | on 28 days
  mortality of patients on 28 days or on a day of discharge if patients are discharged earlier than 28 days
duration of mechanical ventilation | up to 28 days
  duration of mechanical ventilation in the ICU involving non-invasive ventilation

SECONDARY OUTCOMES:
length of stay in the ICU | up to 28 days
length of stay in the hospital | up to 28 days
Evaluation of restlessness and delirium | up to 28 days in the ICU
  evaluation of Richmond agitation-sedation scale (RASS) and Confusion Assessment Method for ICU patients (CAM-ICU)
Evaluation of cognitive function | on 28 days or on the day of discharge
  evaluation of Mini mental state examination (MMSE) on the 28 days or on a day of discharge if patients are discharged earlier than 28 days
Occurrence of arrythmia or myocardial ischemia | up to 28 days in the ICU
Renal function | up to 28 days in the ICU
  blood urea nitrogen (BUN), creatinine, estimated glomerular filtration rate (eGFR), daily urinary output, need of renal replacement therapy
infection control | within 28 days until discharge
  Duration of antimicrobial agents use within 28 days or a day of discharge if patients are discharged earlier than 28 days
inflammation marker | for 14days
  Laboratory marker of inflammation (CRP, PCT) on 1,3,7,14 days
organ failure control | up to 28 days in the ICU
  Sequential Organ Failure Assessment (SOFA) score during in the ICU
coagulopathy control | for 14 days
  Disseminated Intravascular Coagulation (DIC) score by the Japanese Association for Acute Medicine during in the ICU
nutrition control | up to 28 days in the ICU
  daily energy intake by enteral nutrition
sedation control | up to 28 days in the ICU
  dose of sedative drugs and analgesic drugs during in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Yu Kawazoe, Study Chair — Tohoku University; Hitoshi Yamamura, doctor, Study Director — Hirosaki University; Takeshi Morimoto, doctor, Study Director — Hyogo Medical University
Locations (1):
- Tohoku University, Sendai, Miyagi, Japan

REFERENCES:
- [Derived] Ohta Y, Miyamoto K, Kawazoe Y, Yamamura H, Morimoto T. Effect of dexmedetomidine on inflammation in patients with sepsis requiring mechanical ventilation: a sub-analysis of a multicenter randomized clinical trial. Crit Care. 2020 Aug 10;24(1):493. doi: 10.1186/s13054-020-03207-8. PMID 32778146
- [Derived] Nakashima T, Miyamoto K, Shima N, Kato S, Kawazoe Y, Ohta Y, Morimoto T, Yamamura H; DESIRE Trial Investigators. Dexmedetomidine improved renal function in patients with severe sepsis: an exploratory analysis of a randomized controlled trial. J Intensive Care. 2020 Jan 2;8:1. doi: 10.1186/s40560-019-0415-z. eCollection 2020. PMID 31908779
- [Derived] Yamamura H, Kawazoe Y, Miyamoto K, Yamamoto T, Ohta Y, Morimoto T. Effect of norepinephrine dosage on mortality in patients with septic shock. J Intensive Care. 2018 Feb 26;6:12. doi: 10.1186/s40560-018-0280-1. eCollection 2018. PMID 29497535
- [Derived] Kawazoe Y, Miyamoto K, Morimoto T, Yamamoto T, Fuke A, Hashimoto A, Koami H, Beppu S, Katayama Y, Itoh M, Ohta Y, Yamamura H; Dexmedetomidine for Sepsis in Intensive Care Unit Randomized Evaluation (DESIRE) Trial Investigators. Effect of Dexmedetomidine on Mortality and Ventilator-Free Days in Patients Requiring Mechanical Ventilation With Sepsis: A Randomized Clinical Trial. JAMA. 2017 Apr 4;317(13):1321-1328. doi: 10.1001/jama.2017.2088. PMID 28322414
- [Derived] Rudiger A, Singer M. Decatecholaminisation during sepsis. Crit Care. 2016 Oct 4;20(1):309. doi: 10.1186/s13054-016-1488-x. No abstract available. PMID 27716402